CLINICAL TRIAL: NCT04157738
Title: Fixed Dose for Fixed Carbohydrates vs. Variable Dosing for Variable Carbohydrates: A Study of Rapid-Acting Mealtime Insulin in Children and Adolescents With Newly Diagnosed Type 1 Diabetes Mellitus.
Brief Title: A Study of Rapid-Acting Mealtime Insulin in Children and Adolescents With Newly Diagnosed Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Felner, MD, MSCR, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00114078
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes
Keywords: Diabetes; Glycemic variability; Insulin; Parental Stress; Advanced carbohydrates counting; Insulin for meals
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin, Short-Acting; Insulin Lispro; Insulin Aspart; Insulin, Long-Acting; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fixed Group (Experimental): Children and adolescents with newly-diagnosed T1DM will receive a fixed mealtime carbohydrate with a fixed mealtime insulin dose, that is a simplified regimen that provides a set amount of insulin for a set amount of carbohydrates, and ensures that each dose and each meal is consistent.
  Interventions: Drug: Rapid-Acting Insulin; Drug: Long acting insulin
- Insulin to carbohydrate ratio (ICR) Group (Active Comparator): Children and adolescents with newly-diagnosed T1DM will receive an Insulin to carbohydrate ratio (ICR) with variable carbohydrate intake mealtime regimen
  Interventions: Drug: Rapid-Acting Insulin; Drug: Long acting insulin

INTERVENTIONS:
Drug: Rapid-Acting Insulin — Prior to discharge, all subjects will receive a regimen that includes a Meal-time insulin and carbohydrate regimen (number of units of insulin, number of carbohydrates, and/or ICR)
  Other Names: Lispro, Aspart, glulisine
Drug: Long acting insulin — Prior to discharge, all subjects will receive a regimen that includes a daily dose of long-acting insulin (Glargine)
  Other Names: Glargine

SUMMARY:
Type 1 diabetes mellitus (T1DM) is a challenging medical disorder, especially in children and adolescents. In order to prevent the chronic complications of hyperglycemia, the maintenance of near-normal glycemic control must be balanced with minimizing hypoglycemia. Although many pediatric endocrinologists provide an ICR plan for their newly diagnosed patients with T1DM, fixed dosing and other forms of insulin delivery are available. This proposal is designed to compare children and adolescents with newly diagnosed T1DM using a fixed insulin dose for fixed carbohydrate mealtime regimen (FIXED group) to children and adolescents with newly diagnosed T1DM using an ICR with variable carbohydrate intake (ICR group) mealtime regimen. In addition to determining the feasibility for a subsequently larger clinical trial, the aims of this investigator-initiated, prospective proposal, is twofold. The first is to determine if the caregivers of diabetics using a fixed insulin for fixed carbohydrate regimen (FIXED group) experience less anxiety than the caregivers of those using an ICR with variable carbohydrate intake regimen (ICR group) at 1- and 4-months post-randomization. The second is to determine if diabetics utilizing a fixed insulin for fixed carbohydrate regimen (FIXED group) have decreased glycemic variability (GV) than those using an ICR with variable carbohydrate intake regimen (ICR group) at 1- and 4-months post-randomization.

DETAILED DESCRIPTION:
Although children and adolescents with T1DM have much more freedom with the amount of food (carbohydrates) they eat while using an ICR at mealtime, the difficulty in determining the amount of insulin needed, how and when to adjust the ICR, the difficulty with understanding the basics of managing T1DM, and the adaptation to a new lifestyle with T1DM may be more complicated than utilizing a simple plan that includes a fixed amount of insulin and fixed number of carbohydrates, at least for the first few months after diagnosis. As complicated as it is for children, adolescents, and their caregivers to learn how to manage T1DM after being discharged home in usually < 48 hours after diagnosis, a more simplified insulin regimen at mealtime may provide the family of and the child or adolescent with newly diagnosed T1DM with less stress and anxiety while still maintaining adequate glycemic control. Twenty - 40 subjects will be recruited at Children's Hospital of Atlanta (CHOA) at Egleston and will be randomized to either the FIXED group or the ICR group according to a computer-generated random sampling table. The subject and his/her caregivers will receive diabetes education while in the hospital in standard fashion. The subject and his/her caregivers will receive glucose monitoring education and training prior to hospital discharge. The subject and his/her caregivers will also receive a paper log to record the blood sugars, number of carbohydrates consumed and insulin administered at each meal throughout the day.

Prior to discharge, all subjects will receive a regimen that includes a: 1) Meal-time insulin and carbohydrate regimen (# of units of insulin, # of carbohydrates, and/or ICR); 2) Daily dose of Glargine; 3) Hyperglycemia correction regimen for blood glucose levels > 199 mg/dL; and 4) Hypoglycemia treatment regimen for blood glucose levels < 70 mg/dL and/or symptomatic.

As per standard diabetes care, caregivers will report all blood glucose levels every day (to the study investigators) until the subject's initial clinic visit 4-6 weeks after diagnosis. All insulin adjustments will be made by the study investigators.

After the subject's first clinic visit, caregivers will contact the study investigators once a week to report blood glucose levels and the investigators will make adjustments as needed.

All the diabetes clinic visits will occur at the Center for Advanced Pediatrics (CAP), approximately three miles from CHOA-Egleston Hospital. Subjects will attend clinic with one or more of the investigators approximately 1 and 4 months after enrollment.

At each clinic visit, subjects (and their caregivers) will answer standard diabetes questions, subjects will undergo a physical examination, and subjects' objective data (vital signs, glucose meter (GM) data, insulin dosing, and carbohydrate intake) will be collected by the study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Have Confirmed diagnosis of T1DM based on the most recent ADA criteria
* Be 7 - 15 years of age
* Begin monitoring with a glucose monitor prior to discharge from the hospital
* Have the ability to understand and be willing to adhere to the study protocol
* English or Spanish speakers

Exclusion Criteria:

* Have a clinically significant major organ system disease
* Be on glucocorticoid therapy
* Have Type 2 Diabetes Mellitus
* Have Polycystic Ovarian Syndrome (PCOS)
* Have a BMI > 85th %ile
* Have Acanthosis Nigricans
* Have any form of renal impairment
* Have Cystic Fibrosis
* Have Glucocorticoid-, Chemotherapeutic-, or any other Medication-induced form of Diabetes
* Be using any basal insulin other than Glargine insulin
* Have cognitive impairment (> 2 grades behind age-appropriate grade in school)
* Be in Foster Care
* Have any history of Division of Family and Children Services (DFCS) involvement
* If female, be pregnant or breast-feeding.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric I Felner, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz JVR, Figueroa J, Felner EI. A pilot study of mealtime insulin administration and parental stress in youth with new-onset type 1 diabetes. Diabet Med. 2023 Apr;40(4):e15039. doi: 10.1111/dme.15039. Epub 2023 Jan 19. PMID 36617389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Moved out of state | 0 | 2
Not completed — Did not show up to the Follow-up appointment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [9 to 12.5] | 11 [9 to 12] | 11 [9 to 11.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Onset with Acidosis [Count of Participants; unit: Participants]
  Yes | 8 | 8 | 16
  No | 4 | 4 | 8
Pubertal at onset [Count of Participants; unit: Participants]
  Yes | 5 | 5 | 10
  No | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of All Consented Participants
Description: The capacity for recruitment was assessed, including all subjects that signed the Informed Consent Form (ICF).
Time Frame: 4 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

2. Primary Outcome: Number of Participants That Completed All Visits
Description: Number of participants that were able to complete all study visits, including the visits in-person at 1 month and 4 months post-randomization.
Time Frame: 4 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Number analyzed (Participants) | 12 | 12
Participants | 11 | 10

3. Primary Outcome: Caregiver Treatment Adherence at 1 Month and 4 Months Post-intervention
Description: Caregiver treatment adherence was assessed using a blood glucose log. Subjects and caregivers recorded blood glucose levels and the amount/type of insulin given. This data was used to calculate adherence as a percentage ranging from 0% (no adherence) to 100% (full adherence).
Time Frame: 1 month post-intervention and 4 months post-intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Number analyzed (Participants) | 12 | 10
percentage of participants
  < 4 times/day at 1-month visit | 3.2 [0.0 to 16.1] | 10.2 [2.4 to 21.4]
  ≥ 4 times/day at 1-month visit | 96.8 [83.9 to 100] | 89.8 [78.6 to 97.6]
  < 4 times/day at 4-month visit | 2.6 [0.0 to 12.6] | 16.1 [2.0 to 39.2]
  ≥ 4 times/day at 4-month visit | 97.0 [87.4 to 100] | 83.9 [61.8 to 98.0]

4. Secondary Outcome: Caregiver Anxiety
Description: Caregiver anxiety was measured with the "parental stress scale". Caregivers completed the "parental stress scale" at initial enrollment and at each clinic follow up visit. The Parental Stress Scale includes 18 questions that are rated from 1 (strongly disagree) to 5 (strongly agree). Scoring ranges from 18 - 90. The higher the score, the higher the stress and anxiety level.
Time Frame: Baseline, 1 month post-intervention, 4 months post-intervention
Population: Number of participants analyzed include subjects that had visits in-person at 1 month and 4 months post-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 29.1 [24.3 to 34.0] | 30.2 [25.3 to 35.0]
  1 month post-intervention: number analyzed (Participants) | 12 | 9
  1 month post-intervention | 27.0 [22.2 to 31.8] | 35.9 [30.7 to 41.1]
  4 months post-intervention: number analyzed (Participants) | 11 | 10
  4 months post-intervention | 27.6 [22.7 to 32.6] | 34.4 [29.3 to 39.4]

5. Secondary Outcome: Glycemic Variability (GV) at 1 Month and 4 Months Post-intervention
Description: The GV was calculated in all subjects using the average blood glucose levels collected from the daily blood glucose paper log. A subjective qualification system was used to label each subject's GV based on their blood glucose levels and an established glucose monitoring (GM) data system. Subjects are considered to have appropriate GV if their blood glucose levels are in the range of 80 mg/dL - 180 mg/dL. Percentage of participants within each specific average BG range is shown.
Time Frame: 1 month post-intervention, 4 months post-intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
Number analyzed (Participants) | 12 | 10
percentage of participants
  BG < 50 mg/dL at 1 month post-intervention | 0.5 [0.0 to 0.6] | 0.5 [0.0 to 0.7]
  BG 50-79 mg/dL at 1 month post-intervention | 8.9 [4.7 to 14.7] | 8.3 [5.2 to 10.0]
  BG 80-180 mg/dL at 1 month post-intervention | 67.5 [48.9 to 70.0] | 63.2 [54.0 to 74.6]
  BG 181-350 mg/dL at 1 month post-intervention | 25.8 [13.3 to 37.7] | 26.8 [17.1 to 34.0]
  BG >350 mg/dL at 1 month post-intervention | 0.8 [0.0 to 1.6] | 0.3 [0.0 to 2.0]
  BG < 50 mg/dL at 4 month post-intervention | 0.0 [0.0 to 0.2] | 0.4 [0.0 to 1.5]
  BG 50-79 mg/dL at 4 month post-intervention | 8.6 [5.3 to 12.4] | 7.3 [4.2 to 11.4]
  BG 80-180 mg/dL at 4 month post-intervention | 63.3 [57.1 to 80.4] | 69.0 [59.5 to 75.9]
  BG 181-350 mg/dL at 4 month post-intervention | 28.7 [8.2 to 35.5] | 21.8 [5.8 to 28.0]
  BG >350 mg/dL at 4 month post-intervention | 0.1 [0.0 to 0.8] | 0.4 [0.0 to 2.7]

ADVERSE EVENTS:
Time Frame: Data collected during follow up (until 4 months post-intervention).
Arm/Group | Fixed Group | Insulin to Carbohydrate Ratio (ICR) Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Group (N=12) | Insulin to Carbohydrate Ratio (ICR) Group (N=12)
Severe Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Altered Mentas Status (General disorders) | 0 (0) | 0 (0)
Diabetic Keoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04157738/Prot_SAP_000.pdf